CLINICAL TRIAL: NCT03484325
Title: Surgical Joint Registry
Brief Title: Surgical Joint Registry MBJRF
Acronym: MBJRFREG
Status: Enrolling by invitation | Type: Observational
Sponsor: Memorial Bone and Joint Research Foundation (Other)
Responsible Party: Principal Investigator, Stefan Kreuzer MD, President, Memorial Bone and Joint Research Foundation
Other Study IDs: HSC-GEN-09-0143
Record Dates: First submitted 2011-07-22; First posted 2018-03-30 (Actual); Last update posted 2019-08-15 (Actual); Status verified 2019-08

CONDITIONS: Osteoarthritis, Knee; Osteoarthritis, Hip
Keywords: Registry; Joint Registry; OA; Osteoarthritis; Osteo arthritis; knee; hip; tka; tha
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis, Hip; Osteoarthritis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to follow the patient's short term and long term clinical outcome after undergoing joint replacement surgery.

DETAILED DESCRIPTION:
This is a registry database. Consented subjects will have their medical data collected via a patient questionnaire in either paper or web based application form. Data will be collected prospectively and retrospectively and will be entered into the database generated by Memorial Bone and Joint Research Foundation. Collection of data will start during the initial clinic visit as part of standard of care. Subjects will be asked to fill out a 4-page "pre-operative hip questionnaire" or "pre-operative knee questionnaire", which includes questions for self-assessment from the Hip Disability and Osteoarthritis Outcome Score (HOOS), Knee disability and Osteoarthritis Outcome Score (KOOS), EQ-5D and University of California, Los Angeles Activity (UCLA) questionnaires. Demographic, intra-operative and additional data will also be collected to correctly identify the subject's specific disease process and treatment plan. Subjects will be asked to fill out a post-operative hip and knee questionnaire that is similar to the pre-operative questionnaire to evaluate the improvement in their clinical outcomes. The subjects will be requested to complete the post-operative questionnaires at 6 months and annually thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria will be limited to subjects who have consented to undergo elective total joint replacement, hip resurfacing and partial knee surgery, arthroscopy and Femoro-actabular impingement (FAI) release performed by the PI.
* All patients of legal adult age will be eligible for the study. All patients will have an equal chance to participate in the study regardless of race or gender. Patients will be enrolled in the order as they are diagnosed by the PI.

Exclusion Criteria:

* Exclusion criteria will be limited to morbid obesity, active infection, heart failure, lung failure, severe bleeding abnormalities, subject with known metal allergy, subject who cannot legally decide for themselves.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Hip and knee replacement patients treated by the principal investigator.
Sampling Method: Probability Sample
Enrollment: 990 (Estimated)
Dates: Start 2009-05; Primary Completion 2020-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Change of Knee Society Scores with KOOS survey | Pre-operatively (baseline) and at 6 months, 12 months, 24 months, 36 months, 48 months, 60 months, 72 months, 84 months, 96 months, 108 months, 120 months
  The purpose of this study is to follow the patient's short term and long term clinical outcome after undergoing knee replacement surgery.
  These clinical outcomes will be assessed by using the KSS along with the KOOS survey for knee replacement cases. The scores obtained at each time point will be compared to the baseline. Therefore the outcome is the change of scores over time.
Change of Hip Society Scores with HOOS survey | Pre-operatively (baseline) and at 6 months, 12 months, 24 months, 36 months, 48 months, 60 months, 72 months, 84 months, 96 months, 108 months, 120 months
  The purpose of this study is to follow the patient's short term and long term clinical outcome after undergoing hip replacement surgery.
  These clinical outcomes will be assessed by using the HSS for hips along with the HOOS survey for hip replacement cases. The scores obtained at each time point will be compared to the baseline. Therefore the outcome is the change of scores over time.

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Kreuzer, MD, Principal Investigator — Memorial Bone and Joint Research Foundation
Locations (1):
- Memorial Bone & Joint Research Foundation, Houston, Texas, United States